CLINICAL TRIAL: NCT03516045
Title: A Study of 18F-AlF-NOTA-Neurotensin PET/CT for Imaging Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201801002
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
Keywords: 18F-AlF-NOTA-neurotensin
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-AlF-NOTA-neurotensin PET/CT (Experimental): One injection of the radioligand 18F-AlF-NOTA-neurotensin Device: PET/CT Following injection of 18F-AlF-NOTA-neurotensin the participants will be subjected to whole body PET/CT
  Interventions: Drug: 18F-AlF-NOTA-neurotensin

INTERVENTIONS:
Drug: 18F-AlF-NOTA-neurotensin — One injection of the radioligand 18F-AlF-NOTA-neurotensin
  Other Names: 18F-AlF-NOTA-NT

SUMMARY:
The aim of this study is to investigate the clinical value of [18F]aluminum fluoride-1,4,7-triazacyclononane-1,4,7-triacetic acid-neurotensin（18F-AlF-NOTA-neurotensin）positron emission tomography / computed tomography (PET/CT) in patients with prostate cancer (PCa).

DETAILED DESCRIPTION:
18F-AlF-NOTA-neurotensin is a radioligand targeting the neurotensinreceptor, which is widely expressed on the cell surface of PCa. The radioligand can be used for the diagnosis and stage of the PCa. A total of 5 volunteers and 60 PCa patients will be subjected to a 18F-AlF-NOTA-neurotensin PET/CT scan. The uptake of 18F-AlF-NOTA-neurotensin in organs and tumor lesions will be quantified as Standardized Uptake Values (SUVmax/SUVmean).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or clinically confirmed and/or suspicious of PCa.
2. Signed informed consent.

Exclusion Criteria:

Claustrophobia (unable to accept PET/CT scanning)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
18F-AlF-NOTA-neurotensin PET/CT imaging of patients with Prostate Cancer | 12 months
  The radioligand 18F-AlF-NOTA-neurotensin can be used to visualize prostate cancer

SECONDARY OUTCOMES:
18F-AlF-NOTA-neurotensin PET/CT prognostic factor for overall and disease specific survival | 24 months
  The standard uptake value (SUV) of the 18F-AlF-NOTA-neurotensin in prostate cancer lesions is associated with Gleason score, staging and risk stratification of prostate cancer.
  SUV (g/mL)=Cimg / (ID/BW) ; Cimg is the prostate cancer pixel intensities of a calibrated PET image (MBq/ml), ID is the injected dose or injected radioactivity (MBq),BW is the body weight (g) .
  Gleason score of a prostate biopsy or radical prostatectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Yongxiang Tang, MD, Principal Investigator — Department of PET Center,Xiangya Hospital,Central South University
Locations (1):
- Department of PET Center,Xiangya Hospital,Central South University, Changsha, China, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maschauer S, Einsiedel J, Hubner H, Gmeiner P, Prante O. (18)F- and (68)Ga-Labeled Neurotensin Peptides for PET Imaging of Neurotensin Receptor 1. J Med Chem. 2016 Jul 14;59(13):6480-92. doi: 10.1021/acs.jmedchem.6b00675. Epub 2016 Jun 30. PMID 27336295
- [Background] Wu Z, Li L, Liu S, Yakushijin F, Yakushijin K, Horne D, Conti PS, Li Z, Kandeel F, Shively JE. Facile Preparation of a Thiol-Reactive (18)F-Labeling Agent and Synthesis of (18)F-DEG-VS-NT for PET Imaging of a Neurotensin Receptor-Positive Tumor. J Nucl Med. 2014 Jul;55(7):1178-84. doi: 10.2967/jnumed.114.137489. Epub 2014 May 22. PMID 24854793
- [Background] Deng H, Wang H, Wang M, Li Z, Wu Z. Synthesis and Evaluation of 64Cu-DOTA-NT-Cy5.5 as a Dual-Modality PET/Fluorescence Probe to Image Neurotensin Receptor-Positive Tumor. Mol Pharm. 2015 Aug 3;12(8):3054-61. doi: 10.1021/acs.molpharmaceut.5b00325. Epub 2015 Jul 21. PMID 26162008